CLINICAL TRIAL: NCT00614016
Title: A Phase 1, Single-Dose Safety and Pharmacokinetic Study of Sodium ST20 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HemaQuest Pharmaceuticals Inc. (Industry)
Responsible Party: Susan Perrine, MD/ Chief Scientific Officer, HemaQuest Pharmaceuticals, Inc.
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: HQP 2007-001
Record Dates: First submitted 2008-01-18; First posted 2008-02-13 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Healthy
Keywords: healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- single (Experimental): 8 subjects total (6 active and 2 placebo)
  Interventions: Drug: Sodium ST20

INTERVENTIONS:
Drug: Sodium ST20 — single administration of oral dosage form

SUMMARY:
A safety and pharmacokinetic study of a single dose of ST20 in healthy volunteers

DETAILED DESCRIPTION:
A Phase 1 study in healthy volunteers to assess the safety and pharmacokinetics of ST20 after oral administration of a single-dose. In addition, a comparison of the pharmacokinetics and exposure of a single dose of ST20 under fasting and non-fasting conditions will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy male or female
* Be between the ages of 18 and 45 years old, inclusive
* Be able and willing to give informed consent
* Be able to comply with all study procedures
* If female, not be pregnant, including negative serum pregnancy test
* If female, must not be of childbearing potential or must agree to use one or more of the following forms of contraception during screening and throughout the study: hormonal (i.e., oral, transdermal, implant or injection); double barrier (i.e., condom, diaphragm with spermicide); intrauterine device (IUD); vasectomized partner (six months minimum); or abstinence. Male subjects must also agree to use one or more of the above forms of birth control for either themselves or their partner, as appropriate throughout the course of the study
* Must not be receiving prescription medication within the 2 weeks before administration of the test dose, except for multivitamins or contraception
* Have white blood cell count, hemoglobin, hematocrit and platelet count within normal range for the testing facility
* Must have serum chemistry values and urinalysis values within the limits of normal for the testing facility
* Must have coagulation parameters within the limits of normal for the testing facility
* Must have a negative urine test for substances of abuse including marijuana, cocaine, cocaine derivatives, opiates and methadone

Exclusion Criteria:

* Have clinically significant vital signs
* Have any clinically significant laboratory value (CBC, serum chemistry, or urinalysis)
* Have made a blood donation of 500mL within the 2 months before administration of study medication
* Have received a blood transfusion within the 3 months before administration of study medication
* Have an acute febrile illness or upper respiratory tract illness within 72 hours prior to administration of study medication
* Have received another investigational agent within the 4 weeks before administration of test drug
* Have received any other investigational agent during this study
* Have any acute or chronic disease (e.g., history of hepatitis or HIV-1)
* Have cardiac disease including congestive heart failure or arrhythmia
* Have a history of central nervous system disease, such as seizures
* Be breast feeding a child
* Have been a smoker in the past 12 months
* Have Body Mass Index (BMI) > 33 kg/m2

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
safety, maximum tolerated dose | specified timepoints in the protocol

SECONDARY OUTCOMES:
pharmacokinetics | specified timepoints in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Robin Downey, MD, Principal Investigator — Charles River Clinical Services Northwest, Inc.
Locations (1):
- Charles River Clinical Services Northwest, Inc., Tacoma, Washington, United States